CLINICAL TRIAL: NCT01808430
Title: Real World Outcomes of Video-Assisted Thoracoscopic Surgery for Lung Cancer Using ECHELON FLEX™ Powered ENDOPATH® Stapler: a Prospective European Multicenter Study
Brief Title: Powered Echelon Device in VATS Surgery
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CME-12-001
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VATS for NSCLC patients: VATS for confirmed non-small cell lung cancer (NSCLC)
  Interventions: Procedure: VATS for confirmed non-small cell lung cancer (NSCLC)

INTERVENTIONS:
Procedure: VATS for confirmed non-small cell lung cancer (NSCLC) — Video-Assisted Thoracoscopic Surgery for NSCLC patients
  Other Names: Video-Assisted Thoracoscopic Surgery

SUMMARY:
This study aims to collect real world outcomes of Video-Assisted Thoracoscopic Surgery (VATS) for lung cancer (lobectomy, wedge resection) using ECHELON FLEX™ Powered ENDOPATH® Staplers 45 mm and/or 60 mm (study devices).

DETAILED DESCRIPTION:
The European prospective observational multi-center cohort study aims to collect real-world outcomes of consecutive patients scheduled for VATS lobectomy for histologically confirmed Non-Small Cell Lung Cancer (NSCLC) or scheduled for VATS wedge resection for undiagnosed pulmonary nodule or metastasis from colorectal cancer (CRC) in accordance with their institution's Standard-of-care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (up to and including Stage II) for patients undergoing VATS lobectomy. For patients undergoing wedge resection for undiagnosed pulmonary nodule or metastasis from CRC, a malignant diagnosis may be confirmed post-operatively.
* Scheduled for lung resection surgery (lobectomy or wedge resection) involving only one lobe of the lung
* Willing to give consent and comply with evaluation and treatment schedule
* At least 18 years of age

Exclusion Criteria:

* Active bacterial infection or fungal infection
* Systemic administration (intravenous or oral) of steroids (within 30 days prior to study procedure)
* Chemotherapy or radiation therapy for lung cancer may not be performed for 30 days prior to the procedure
* Scheduled concurrent surgical procedure other than wedge resection or lobectomy (central venous access - e.g. port placement, mediastinoscopy with lymph node sampling, and VATS lymphadenectomy are allowed);
* Prior history of VATS or open lung surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for VATS lobectomy for histologically confirmed Non-Small Cell Lung Cancer (NSCLC) or scheduled for VATS wedge resection for undiagnosed pulmonary nodule or metastasis from colorectal cancer (CRC) in accordance with their institution's Standard-of-care (SOC).
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
occurrence and duration of post-operative air leak | prolonged air leak defined as longer than 5 days post-op
  occurrence and duration of prolonged air leak defined as longer than 5 days

SECONDARY OUTCOMES:
volume of estimated intra-operative blood loss | blood loss intra-op and up to 5 days post-op
  volume of estimated intra-operative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ribaric, MD, MSc, PhD, Study Chair — Ethicon Endo-Surgery (Europe) GmbH
Locations (1):
- Professor Peter Licht, Odense, Denmark